CLINICAL TRIAL: NCT05049993
Title: Pyrocarbon Clinical Follow-up Study
Acronym: PYC CFS
Status: Active, not recruiting | Type: Observational
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: 20A-W-PYC-RM
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Osteoarthritis of the Shoulder; Avascular Necrosis; Traumatic Arthritis
MeSH Terms: conditions — Osteonecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Aequalis Pyrocarbon Humeral Head — Hemi Shoulder Arthroplasty using the Aequalis Pyrocarbon Humeral Head

SUMMARY:
The objective of this multi-center study is to collect medium and long-term data on the related clinical complications and functional outcomes of the Pyrocarbon Humeral Head to demonstrate safety and performance, in subjects from the Pyrocarbon IDE Study cohort.

Data collected from this study will support post-market surveillance and MDR requirements as well provide the basis for peer-reviewed publications on mid- and long-term product performance and safety (five to ten years post-op).

ELIGIBILITY:
Inclusion Criteria:

* Subject in the Pyrocarbon IDE Study and has not had the device explanted.
* Patient informed, willing, and able to sign an informed consent form approved by IRB or EC
* Willing and able to comply with the requirements of the study protocol

Exclusion Criteria:

• Subjects who are not able to comply with the study procedures based on the judgment of the assessor will be excluded (e.g. cannot comprehend study questions, inability to keep scheduled assessment times)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Long-term follow-up of Pyrocarbon IDE patients.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to last follow-up visit in ASES scores | Follow-up visits through 10 years Post-Op
  ASES Score = American Shoulder and Elbow Surgeons Score, 11 items with total score reported out of 100 measuring pain and activity of patient's evaluated shoulder where lower scores indicate more pain and less function

SECONDARY OUTCOMES:
Change from Baseline to last follow-up visit in Constant Murley scores | Follow-up visits through 10 years Post-Op
  Combination of physician-completed and patient-reported portions to assess functional state of shoulder including range of motion; total score reported out of 100 measuring where lower scores indicate less function of the evaluated shoulder
Change from Baseline to last follow-up visit in SANE scores | Follow-up visits through 10 years Post-Op
  SANE = Single Assessment Numeric Evaluation; 1 item assessment of shoulder rating 0% to 100%
Change from Baseline to last follow-up visit in Subject Satisfaction scores | Follow-up visits through 10 years Post-Op
  Single, subjective question measuring patient satisfaction; assessed by improved, worsened, or no change in satisfaction
Change from Baseline to last follow-up visit in EQ-5D scores | Follow-up visits through 10 years Post-Op
  The EuroQol Five Dimensions Questionnaire (EQ-5D) questionnaire is a standardized instrument for use as a measure of quality of life. It is cognitively simple, takes only a few minutes to complete, and provides a simple descriptive profile as well as a single index value for quality of life that can be used in the clinical and economic evaluation of health care. The EQ-5D consists of a descriptive system which comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression), and a visual analog scale which measures the respondent's self-rated health on a 0-100 scale.
Number of device associated and procedure associated adverse events. | Follow-up visits through 10 years Post-Op
Evaluation of operated shoulder range of motion | Follow-up visits through 10 years Post-Op
Rates of revision surgeries. | Follow-up visits through 10 years Post-Op

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gibson, Study Director — Stryker Trauma & Extremities
Locations (8):
- United States (8):
  - HCA HealthONE, LLC, Denver, Colorado
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Tulane University, New Orleans, Louisiana
  - Southern Maryland Orthopedics, Waldorf, Maryland
  - Allina Health Orthopedics, Minneapolis, Minnesota
  - Missouri Orthopaedic Institute, Columbia, Missouri
  - Duke University, Durham, North Carolina
  - Southern Oregon Orthopedics, Medford, Oregon

IPD SHARING:
Plan to Share IPD: No